CLINICAL TRIAL: NCT04719195
Title: Comparison of Meniscus Extrusion Between Preoperative and Postoperative Medial Opening Wedge High Tibial Osteotomy by Using Ultrasonographic Assessment
Brief Title: Comparison of Meniscus Extrusion Between Preoperative and Postoperative MOWHTO Using Ultrasonographic Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Other Study IDs: KC20OISI0561
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Meniscus extrusion ultrasonogrphic evaluation — This study will enroll the patients with knee medial compartment osteoarthritis of the knee joint who undergo open proximal tibial osteotomy. The degree of medial and lateral meniscus extrusion will be measured through ultrasound measurements before and after surgery. Also, demographic factors and radiographic measurements will be also investigated before and after surgery. In addition, preoperative, postoperative 3, 6, and 1 year clinical results including meniscus extrusion will be compared and judged, and the evaluation will be evaluated by an orthopedic surgeon who has not participated in the operation among registered researchers.

SUMMARY:
The purpose of this study is to measure the changes in the medial and lateral meniscus extrusion of the knee joint before and after surgery using ultrasound in patients who undergo medial opening wedge high tibial osteotomy, and examine the differences.

DETAILED DESCRIPTION:
High tibial osteotomy (HTO) is an established treatment method for medial compartment osteoarthritis with varus knee deformity in a relatively young patient group. Excellent outcomes of HTO have been reported. However, about 10-30% of patients are not satisfied with the results after surgery. After proximal tibial osteotomy, studies on the factors of dissatisfaction have been actively conducted, but studies on the medial and lateral meniscus extrusion, which can be the cause, are insufficient. The relationship between the prolapse of the medial meniscus and articular cartilage is already well known and is known as an important factor in the progression of arthritis. As such, the association between the knee joint with meniscus extrusion and the general knee joint has been studied, but the effect on the clinical outcome after proximal tibial osteotomy has not been studied. Therefore, in this study, the investigators are planning to investigate the differences in clinical outcomes such as the degree and change of medial and lateral meniscus extrusion through non-invasive ultrasound examination before and after surgery in patients who undergo medial open proximal tibial osteotomy.

This study will enroll the patients with knee medial compartment osteoarthritis of the knee joint who undergo open proximal tibial osteotomy. The degree of medial and lateral meniscus extrusion will be measured through ultrasound measurements before and after surgery. Also, demographic factors and radiographic measurements will be also investigated before and after surgery. In addition, preoperative, postoperative 3, 6, and 1 year clinical results including meniscus extrusion will be compared and judged, and the evaluation will be evaluated by an orthopedic surgeon who has not participated in the operation among registered researchers.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20
* Medial compartment knee osteoarthritis patients for Medial Opening Wedge High Tibial Osteotomy
* Patients who are willing or able to follow doctor's instructions, including joint exercises
* Patients who have received sufficient explanation for this clinical trial and agreed to participate

Exclusion Criteria:

* Patients with secondary knee osteoarthritis
* Patients with inflammatory arthritis or crystalline arthritis
* Local infection to the lower extremities of the pain area, sepsis, or previous neurological abnormalities.
* Patients with knee range of motion less than 90 degrees
* Patients with BMI above 40

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medial compartment knee osteoarthritis patients for Medial Opening Wedge High Tibial Osteotomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2022-07-24 (Estimated); Study Completion 2022-07-24 (Estimated)

PRIMARY OUTCOMES:
WOMAC(Western Ontario and McMaster University Arthritis Index ) pain scale | changes from pre-operative WOMAC score at post-operative 3rd month, 6th month and 1 year

SECONDARY OUTCOMES:
Pain Visual Analogue Scale | changes from pre-operative VAS score at post-operative 3rd month, 6th month and 1 year
SF-12(Short Form heath survey) score | changes from pre-operative SF-12 score at post-operative 3rd month, 6th month and 1 year
EQ-5D(EuroQoL-5 Dimension) | changes from pre-operative EQ-5D score at post-operative 3rd month, 6th month and 1 year
X-ray | changes from pre-operative Kellgren-Lawrence grade at post-operative 3rd month, 6th month and 1 year
  Kellgren-Lawrence grade
X-ray | changes from pre-operative weight bearing line ratio at post-operative 3rd month, 6th month and 1 year
  weight bearing line ratio
Knee range of motion | changes from pre-operative knee range of motion at post-operative 3rd month, 6th month and 1 year
Ultrasonographic evaluation of medial and lateral meniscus extrusion | changes from pre-operative ultrasonographic evaluation of medial and lateral meniscus extrusion at post-operative 3rd month, 6th month and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- the Catholic Univerisity of Korea Seoul St Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No